CLINICAL TRIAL: NCT01329653
Title: Exercise, Age-Related Memory Decline, And Hippocampal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Richard Sloan, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: #6219/#7161R; AG035015 (Other: CU)
Record Dates: First submitted 2010-07-28; First posted 2011-04-06 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cognitive Deterioration; Disorder of Aging
Keywords: cerebral blood volume; aging; exercise
MeSH Terms: conditions — Motor Activity | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aerobic training (Experimental): 12 weeks of aerobic training, 4X/week
  Interventions: Behavioral: aerobic training
- wait list control (Placebo Comparator): wait list control condition, 12 weeks to parallel the active intervention group
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: aerobic training — 12 weeks of aerobic training, 4X/week
  Arms: aerobic training
Behavioral: Wait list — wait list control condition
  Other Names: Wait list control
  Arms: wait list control

SUMMARY:
The purpose of this study is to test the hypothesis that aerobic exercise leads increased cerebral blood volume in the dentate gyrus of the hippocampus in a sample of young and older adults.

DETAILED DESCRIPTION:
In the US, increased length of life and reduced morbidity and mortality have resulted in a growing number of older adults, the demographic "time bomb" often referred to in discussions of public policy. According to the Census Bureau, the population aged 65 and over will double in size within the next 25 years. Moreover, these older adults will live healthier lives than their predecessors. While this increased length of a healthy life is an undeniable societal benefit, it brings with it a major societal problem: an epidemic of aging-related cognitive decline. The need to develop interventions to address this growing problem is urgent. Aging-related cognitive dysfunction is not diffuse; rather it targets selected brain areas, in particular the frontal lobes and the hippocampal formation. The separate but interconnected subregions of the hippocampus are differentially vulnerable to pathogenic mechanisms, including the normal aging process. A range of in vivo and post-mortem studies have converged on the dentate gyrus (DG) as the hippocampal subregion differentially targeted by the aging process. As with pathogenic processes, any intervention that improves brain function does so with regional selectivity. One such intervention is physical exercise, which has been shown to improve both frontal lobe and hippocampal function. Using a high-resolution variant of functional magnetic resonance imaging (fMRI), the investigators have demonstrated that aerobic training selectively benefitted DG function both humans and mice. In addition, improvement in DG function was associated with improved performance on a word list learning task but not in tasks conventionally thought to be frontal lobe dependent. The human part of the study had significant shortcomings, however: it was small (N = 11), lacked a control group, enrolled only young subjects (age 20-45 years), and employed only a limited neuropsychological testing battery. The overall goal of this proposal is to use the high-resolution variant of fMRI to test the hypothesis that aerobic training will induce improvements in DG function in a sample of younger (age 20-35) and older (50-65) adults, assigned randomly to an active training condition or wait list control group. The investigators will use more comprehensive neuropsychological testing to examine the relationship between changes in DG function and selected cognitive capacities. Taken together with the observation that normal aging differentially targets the DG, this research program will establish that physical exercise is an effective approach for ameliorating the insidious cognitive slide that occurs in aging. Thus, the potential significance of this application is substantial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-75 years
2. English-speaking
3. Ambulatory
4. "Average" fitness as determined by ACSM's Guidelines for Exercise Testing and Prescription (for men, VO2max < 43 for age 20-39 years, < 38 for age 40-49 years, < 35 for age 50-59, < 31 for age 60-75; for women, < 36 for age < 30 years, < 34 for age 30-39 years, < 32 for age 40-49 years, <25 for age 50-59 years, < 24 for age 60-75 years
5. BMI <35

Exclusion Criteria:

1. Ischemic changes or abnormal resting cardiogram, abnormal blood pressure responses, or an significant ectopy during aerobic capacity testing
2. Cardiovascular disease
3. BMI > 35
4. Uncontrolled high blood pressure (systolic blood pressure ≥ 140 mmHg; or diastolic blood pressure ≥ 90mmHg on two measures)
5. Any condition for which aerobic training is counter-indicated, including persons with evidence or history of medical or orthopedic conditions which might make participation problematic.
6. Current or recent (evidence of disease x 5 years) non-skin neoplastic disease or melanoma. Prostatic carcinoma will not be grounds for exclusion.
7. Active hepatic disease (not a history of hepatitis) or primary renal disease requiring dialysis, primary untreated endocrine diseases, e.g., Cushing's disease or primary hypothalamic failure or insulin dependent diabetes (Type I or II). Welltreated hypothyroidism will not be excluded.
8. History of chemotherapy
9. HIV infection
10. Pregnant or lactating (participation allowed 3 months after ceasing lactation).
11. Medications that alter inflammation or autonomic nervous system activity
12. Any history of psychosis or ECT
13. Current or recent (past one year) Major Depressive Disorder, Bipolar Disorder
14. Current or recent (within past 12 months) alcohol or substance abuse or dependence. Recent use (past month) of recreational drugs.
15. Dementia Rating Scale (DRS) score less than 135. Medical History Interview
16. Neurological Disorders Dementia Rating Scale
17. Stroke Telephone screen
18. Alzheimer's Disease Telephone screen
19. Smoking Telephone screen
20. Prior participation in another Dr. Sloan Exercise Study
21. MRI Exclusion Criteria: Cardiac Pacemaker; Internal Pump; Insulin Pump; Tattoo; eyeliner; Wire Sutures; Internal Metal Objects; Metal Slivers in Eye; Prosthesis; Hearing Aid Implants; Neurostimulator; Metal Fragments; Brain Aneurysm Clips; Vascular Clips; Breast Expander; Vena Cava Filter; Heart Valve; Metal Stents; Asthma; Hay-Fever; Sickle Cell Disease; Kidney Disease; Machinist or ever worked with heavy metals Interview; Contraindication to gadolinium, including prior adverse reaction to gadolinium, past or current history of severe breathing difficulty that has been treated by a physician (e.g., asthma, COPD, etc.), and sickle cell disease. History of renal impairment or estimated glomerular filtration rate <30 L/min/1.73m2 is also exclusionary; Machinist or ever worked with heavy metals Interview; Have had more than one MRI scans with Gadolinium

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
dentate gyrus cerebral blood volume | change from before (pre) to after (post) 12 weeks of training

SECONDARY OUTCOMES:
cognitive function | change from before (pre) to after (post) 12 weeks of training
  measures of memory, executive function, attention/processing speed, language, and general intelligence
aerobic capacity | change from before (pre) to after (post) 12 weeks of training
cerebral blood flow | change from before (pre) to after (post) 12 weeks of training
  arterial spin labeling fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Sloan, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share our data with other investigators upon request.

REFERENCES:
- [Result] Pereira AC, Huddleston DE, Brickman AM, Sosunov AA, Hen R, McKhann GM, Sloan R, Gage FH, Brown TR, Small SA. An in vivo correlate of exercise-induced neurogenesis in the adult dentate gyrus. Proc Natl Acad Sci U S A. 2007 Mar 27;104(13):5638-43. doi: 10.1073/pnas.0611721104. Epub 2007 Mar 20. PMID 17374720